CLINICAL TRIAL: NCT03889067
Title: Exploring the Bottleneck Hypothesis of the Pathogenesis of Bacteraemia in an Ambulatory Outpatient Human Experimental Infection of Salmonella Typhi
Brief Title: Understanding How Salmonella Typhi Infects Humans (Bottlenecks)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OVG/2018/06
Record Dates: First submitted 2019-03-05; First posted 2019-03-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2020-02

CONDITIONS: Salmonella Typhi Infection
Keywords: Enteric fever; Typhoid; Salmonella Typhi; Typhoid fever; Salmonella infections; Gram-negative bacterial infections; Human model of infection
MeSH Terms: conditions — Typhoid Fever; Salmonella Infections; Gram-Negative Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Ambulatory outpatient human experimental infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Challenge Agents (Experimental): Wild-Type Quailes Strain Salmonella Typhi: Quailes Typhoid toxin knock out strain in a 1:1 ratio at a dose of 1-5 x 10^4CFU
  All participants will receive the same intervention in a given group for challenge (dose reduction may occur for later participants depending on the results from the first six participants)
  Interventions: Biological: Salmonella Typhi challenge

INTERVENTIONS:
Biological: Salmonella Typhi challenge — The challenge agents will be delivered in 30 ml of sodium bicarbonate solution, preceded by 120 ml of solution of sodium bicarbonate to neutralise gastric acid.

SUMMARY:
Typhoid fever is an infection caused by the bacteria Salmonella Typhi (S. Typhi). S. Typhi causes disease principally in developing countries where communities do not have access to safe water or adequate sanitation. It is thought to cause illness in approximately 22 million people every year and up to 200,000 deaths, mostly in children. The bacteria are spread when faeces from infected individuals contaminate food and water sources. Symptoms of infection include headache, fever and general aches and pains. If not treated properly typhoid infection can lead to severe complications and even death.

In this study the investigators aim to understand more about the S. Typhi bacteria and how S. Typhi causes a bloodstream infection after it has been ingested and passed into the gut. In spite of the extensive morbidity and mortality associated with bacterial blood stream infections (BSI), comparatively little is known about the pathogenesis. At a time of increasing antimicrobial resistance and a lack of new antimicrobial agents, understanding the pathogenesis of BSI is essential for efforts directed at prevention both of Salmonella Typhi and other bacterial species, particularly those that are restricted to humans.

DETAILED DESCRIPTION:
The pathogenesis of bacteraemia for human restricted pathogens such as Streptococcus pneumoniae, Haemophilus influenzae type b and Salmonella enterica serovar Typhi (ST), have thus far only been investigated in imperfect animal models. The Salmonella Typhimurium mouse model is widely employed however there are key differences compared with S. Typhi. These bacteria are both genetically distinct and cause a different human disease phenotype . Data from a human model would be invaluable in furthering our understanding of bacteraemia in the human host. Animal studies with Salmonella species and other bacterial species show some evidence that there may be population bottlenecks in the development of blood stream infections.

Inoculation with many microorganisms is often sufficient to cause a blood stream infection in a susceptible host, typically inoculation with a single microorganism is not. There are two principle theories as to how bacteraemia arises. The first is independent action whereby the bacteraemia that results from bacterial inoculation is derived from a single founder organism ('the bottleneck hypothesis'). Each organism has a chance of being that founder organism. A greater number of organisms make bacteraemia more likely. The second theory is synergy where there is cooperation between bacteria, multiple bacteria traverse the barrier to infection and therefore the bacteraemia is composed of multiple variants.

The aim of this research project is to investigate the population bottleneck theory in the pathogenesis of bacteraemia in human infection model using a challenge combination of two isogenic strains of S. Typhi.

The primary objective of the study is to compare the number of participants who develop bacteraemia post challenge from each S. Typhi variant or a combination of the two strains. From animal models the investigators hypothesize that in an individual participant a single strain will be isolated more commonly than a combination of the two. The secondary objectives are to quantify the burden of bacteraemia of the two strains and to characterise the stool shedding in participants given a mixed inoculum.

Exploratory objectives include comparison of the number of participants who develop bacteraemia at various timepoints until 72 hours from each S. Typhi variant or a combination of the two strains. From animal models it is expected that any so-called 'primary bacteraemias' may involve a combination of the S. Typhi strains. The researchers also anticipate that stool cultures from study participants may culture a combination of the S. Typhi strains initially but that if a single isolate is cultured from the blood that this will be reflected in stool culture. The investigators will explore if quantitation of S. Typhi is possible in stool. They will also seek to evaluate the host immune response to challenge in terms of cytokine and blood transcriptional signatures.

This is the first time in which the bottleneck theory has been explored in a human model of a bloodstream infection. It will not only be significant for understanding the pathogenesis of S. Typhi but also for other bacterial pathogens. If this hypothesis is supported this implies that the barrier for vaccine prevention of bacterial infection may be lower than previously thought, perhaps only very few or even a single organism must be prevented from invasion to provide individual protection.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy all of the following criteria to be considered eligible for the study:

  * Agree to give informed consent for participation in the study.
  * Aged between 18 and 60 years inclusive at time of challenge.
  * In good health as determined by medical history, physical examination and clinical judgment of the study team.
  * Agree (in the study team's opinion) to comply with all study requirements, including capacity to adhere to good personal hygiene and infection control precautions.
  * Agree to allow his or her GP (General Practitioner) (and/or Consultant if appropriate), to be notified of participation in the study.
  * Agree to allow study staff to contact his or her GP to access the participant's medical history and vaccination records.
  * Agree to allow Public Health England to be informed of their participation in the study.
  * Agree to give his or her close contacts written information informing them of the participant's involvement in the study and offer them voluntary screening for S. Typhi carriage.
  * Agree to have 24-hour contact with study staff during the four weeks post challenge and are able to ensure that they are contactable by mobile phone for the duration of the challenge period until antibiotic completion.
  * Agree to allow the study team to hold the name and 24-hour contact number of a close friend, relative or housemate who will be kept informed of the study participant's whereabouts for the duration of the challenge period (from the time of challenge until completion of antibiotic course). This person will be contacted if study staff are unable to contact the participant.
  * Have internet access on a daily basis to allow completion of the e-diary and real-time safety monitoring.
  * Agree to avoid antipyretic/anti-inflammatory treatment from the time of challenge (Day 0) until advised by a study doctor or until 14 days after challenge.
  * Agree to refrain from donating blood for the duration of the study
  * Agree to provide their National Insurance/Passport number for the purposes of TOPS (The Over volunteering Prevention System) registration and for payment of reimbursement expenses.
  * Agree not to take part in another research study involving an IMP (Investigational Medicinal Product) or challenge for the entire period of recruitment in the current study.

Exclusion Criteria:

The participant will not be enrolled if any of the following apply:

* History of significant organ/system disease that could interfere with trial conduct or completion. Including, for example, but not restricted to:

  * Cardiovascular disease
  * Respiratory disease
  * Haematological disease
  * Endocrine disorders
  * Renal or bladder disease, including history of renal calculi
  * Biliary tract disease, including biliary colic, asymptomatic gallstones or previous cholecystectomy
  * Gastro-intestinal disease including requirement for antacids, H2-receptor antagonists, proton pump inhibitors or laxatives
  * Neurological disease
  * Metabolic disease
  * Autoimmune disease
  * Psychiatric illness requiring hospitalisation or known or suspected current drug and/or alcohol misuse (alcohol misuse defined as an intake exceeding 42 units per week)
  * Infectious disease
* Have any known or suspected impairment of immune function, alteration of immune function, or prior immune exposure that may alter immune function to typhoid resulting from, for example:

  * Congenital or acquired immunodeficiency, including Immunoglobulin A deficiency
  * Human Immunodeficiency Virus infection or symptoms/signs suggestive of an HIV-associated condition
  * Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 12 months or long-term systemic corticosteroid therapy
  * Receipt of immunoglobulin or any blood product transfusion within 3 months of study start.
  * History of cancer (except squamous cell or basal cell carcinoma of the skin and cervical carcinoma in situ).
* Screening positive for HLA B27 gene.
* Moderate or severe depression or anxiety as classified by the Hospital Anxiety and Depression Score (score 11 or higher on either score) at screening or before challenge that is deemed clinically significant by the study doctors .
* Weight less than 50kg .
* Presence of implants or prosthetic material.
* Anyone taking long-term medication (e.g. analgesia, anti-inflammatories or antibiotics) that may affect symptom reporting or interpretation of the study results.
* Contraindication to ciprofloxacin or macrolide antibiotics.
* Female participants who are pregnant, lactating or who are unwilling to ensure that they or their partner use effective contraception 30 days prior to enrolment/challenge and continue to do so until three negative stool samples, the first taken a minimum of 1 week after completion of antibiotic treatment and subsequent samples at least 48 hours apart each have been obtained.
* Occupational (unless willing and able to confirm that they are not working in the following environment for the period of challenge to clearance confirmation):

  * Full-time, part-time or voluntary occupations involving:

    * Clinical or social work with direct contact with young children (defined as those attending pre-school groups or nursery or aged under 2 years), or
    * Clinical or social work with direct contact with highly susceptible patients or persons in whom typhoid infection would have particularly serious consequences (unless willing to avoid work for at least 6 weeks until demonstrated not to be infected with S. Typhi in accordance with guidance from Public Health England and willing to allow study staff to inform their employer).
  * Full time, part time or voluntary occupations involving:

    * Commercial food handling (involving preparing or serving unwrapped foods not subjected to further heating)
* Close household contact with:

  * Young children (defined as those attending pre-school groups, nursery or those aged less than 2 years)
  * Individual(s) who is (are) immunocompromised.
* Scheduled elective surgery (including dental work) or other procedures requiring general anaesthesia during the study period.
* Participants who have participated in another research study involving an investigational product that might affect risk of typhoid infection or compromise the integrity of the study within the 30 days prior to enrolment (e.g. significant volumes of blood already taken in previous study) .
* Detection of any abnormal results from screening investigations (at the clinical discretion of the study team).
* Inability to comply with any of the study requirements (at the discretion of the study staff and the participant's General Practitioner).
* Any other social, psychological or health issues which, in the opinion of the study staff, may

  * Put the participant or their contacts at risk because of participation in the study,
  * Adversely affect the interpretation of the primary endpoint data,
  * Impair the participant's ability to participate in the study.
* Having previously received any typhoid vaccine within the last 3 years.
* Having been resident in an enteric fever endemic country for 6 months or more .
* Have previously been diagnosed with laboratory-confirmed typhoid or paratyphoid infection or been given a diagnosis compatible with enteric fever.
* Have participated in previous typhoid or paratyphoid challenge studies (with ingestion of challenge agent).
* Have a prolonged corrected QT interval (>450 milliseconds) on ECG screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with a bacteraemia | Two weeks after typhoid challenge
  Number of participants with a bacteraemia caused by wild-type S. Typhi or Typhoid toxin knock-out strain or a combination of both strains as assessed by identification of strains isolated from blood cultures

SECONDARY OUTCOMES:
Number of isolates that are wild-type S.Typhi or Typhoid toxin knock-out strain | Two months after typhoid challenge
  Number of isolates that are wild-type S.Typhi or Typhoid toxin knock-out strain obtained using quantitative blood cultures
umber of participants with positive stool cultures caused by wild-type S. Typhi or Typhoid toxin knock-out strain or a combination of both strains | Six weeks after typhoid challenge
  Number of participants with positive stool cultures caused by wild-type S. Typhi or Typhoid toxin knock-out strain or a combination of both strains as assessed by identification of strains isolated from stool cultures

OTHER OUTCOMES:
Number of participants with a bacteraemia caused by wild-type S. Typhi or Typhoid toxin knock-out strain or a combination of both strains | Two weeks after typhoid challenge
  Number of participants with a bacteraemia caused by wild-type S. Typhi or Typhoid toxin knock-out strain or a combination of both strains as assessed by identification of strains isolated from blood cultures (obtained at less than 72 hours post challenge)
Proportion of stool culture isolates are wild-type S.Typhi or Typhoid toxin knock-out strain | Six weeks after typhoid challenge
  To count what proportion of stool culture isolates are wild-type S.Typhi or Typhoid toxin knock-out strain obtained using quantitative stool cultures
Number of responses obtained from each recruitment method used and number of responses which translated into participants. Number of participants excluded and reasons for exclusion. | 4 weeks after typhoid challenge
  Number of responses obtained from each recruitment method used and number of responses which translated into participants. Number of participants excluded and reasons for exclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, FRCPCH, PhD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Direct access will be granted to authorised representatives from the Sponsor and host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections.